CLINICAL TRIAL: NCT02489747
Title: Efficacy and Safety of Wheat Bran Extract on Improvement of Cognitive and Memory Function
Brief Title: Effects of Wheat Bran Extract on Cognitive and Memory Function
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chonbuk National University Hospital (Other)
Responsible Party: Principal Investigator, Soo-Wan Chae, Professor, Chonbuk National University Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: CTCF2_2013_WBE
Record Dates: First submitted 2015-06-30; First posted 2015-07-03 (Estimated); Last update posted 2016-03-15 (Estimated); Status verified 2016-03

CONDITIONS: Cognitive Function 1, Social
Keywords: cognitive function; CNT; memory function; Triticum aestivum L; wheat bran

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- WBE group (Experimental): wheat bran extract
  Interventions: Dietary Supplement: WBE
- Placebo group (Placebo Comparator): placebo
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: WBE — wheat bran extract (3 g/day)
  Arms: WBE group
Dietary Supplement: Placebo — Placebo
  Arms: Placebo group

SUMMARY:
The investigators performed a 12-week, randomized, double-blind, placebo-controlled human trial to evaluate the efficacy and safety of water extract from wheat Triticum aestivum L on cognitive and memory function. The investigators measured changes in cognitive function parameters, including CNT, WMT, K-MMSE, BCRS, PRMQ, PSS, SF-36 and BDNF

DETAILED DESCRIPTION:
Based on reports about the neuroprotective effects of water extract from wheat Triticum aestivum L. or its bran, the investigators hypothesize that extract of wheat bran (WBE) is beneficial to elderly people with age-associated cognitive impairment. The investigators investigated the efficacy and safety of WBE on improvement of cognitive function through measuring the neuropsychometric assessments in adult with subjective cognitive impairment by a randomized clinical trial.

Seventy participants aged from 50 to 80 years old with subjective cognitive impairment were randomly assigned to receive either WBE (3,000 mg/day) in this 12-week, double-blind placebo-controlled and parallel trial. Neuropsychological assessments including Computerized Neurocognitive function test (CNT), Working Memory Test (WMT), Korean Mini-Mental State Examination (K-MMSE), Brief Cognitive Rating Scale (BCRS), Prospective and Retrospective Memory Questionnaire (PRMQ), Perceived Stress Scale (PSS), 36-Item of Short-Form Health Survey (SF-36) and blood Brain-derived neurotrophic factor (BDNF) were used to assess the cognitive function before and after the intervention.

ELIGIBILITY:
Inclusion Criteria:

* subjects with subjective cognitive impairment
* able to give informed consent

Exclusion Criteria:

* history of underlying neurodegenerative disease
* allergic or hypersensitive to any of the ingredients in the test products
* history of reaction to any of the test products or of gastrointestinal diseases such as Crohn's disease or gastrointestinal surgery
* history of alcohol or substance abuse
* participation in any other clinical trials within past 2 months
* laboratory test, medical or psychological conditions deemed by the investigators to interfere with successful participation in the study etc.

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2013-11; Primary Completion 2014-09 (Actual); Study Completion 2015-02 (Actual)

PRIMARY OUTCOMES:
Cognitive function as assessed by the visual learning test score of CNT (computerized neurocognitive test) | baseline and 12 weeks

SECONDARY OUTCOMES:
Visual subset of WMT (working memory test) | baseline and 12 weeks
Cognitive function as assessed by the CNT (Computerized Neurocognitive Test) score | baseline and 12 weeks
Cognitive function as assessed by the Verbal subtest of WMT (Working Memory Test) | baseline and 12 weeks
Cognitive function as assessed by the BCRS (Brief Cognitive Rating Sclae) | baseline and 12 weeks
Memory function as assessed by the PRMQ (Prospective and Retrospective Memory Questionnaire) | baseline and 12 weeks
Stress level evaluation as assessed by the Perceived stress scale (PSS) | baseline and 12 weeks
Quality of life as assessed by the 36-item short-form healthy survey (SF-36) score | baseline and 12 weeks
Cognitive function as assessed by the Brain-Derived Neurotrophic Factor (BDNF) | baseline and 12 weeks